CLINICAL TRIAL: NCT05263414
Title: Modulation of Neurocognitive Mechanisms Involved in Inhibitory Control in Tic Disorders
Brief Title: Neuromodulation of Inhibitory Control in Tic Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 847
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Tic Disorders
Keywords: Transcutaneous vagus nerve stimulation; Tic disorders; Tourette syndrome; Inhibition; Tic control
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome; Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Active Comparator): In the active tVNS session, tVNS will be delivered via a programmable stimulation unit connected to two titan ear electrodes mounted on a gel frame. Active tVNS will be delivered over the cymba conchae of the left ear for a 70 minutes session. Stimulation intensity will be set at an intensity corresponding to individual sensitivity threshold. The intensity of the stimulation will be gradually increased in order to reach the intensity of stimulation with a ramping-up phase of 30 secs. During the stimulation, participants will perform the tasks. At the end of the stimulation session participants will be asked to report possible side effects occurring during tVNS and to rate their feeling on several visual analogue scales.
  Interventions: Device: tVNS
- Sham tVNS (Sham Comparator): In the sham tVNS session tVNS will be delivered via a programmable stimulation unit connected to two titan ear electrodes mounted on a gel frame. Sham tVNS will be delivered over the left lobe auricle area, which is free from cutaneous vagal innervation. It will last 70 minutes. Stimulation intensity will be set at the intensity corresponding to the individual sensitivity threshold, as it will be defined on the left ear lobe. The intensity of the stimulation will be gradually increased to reach the intensity of the stimulation with a ramping up phase of 30 secs. During the sham stimulation, the tasks will be performed. At the end of the stimulation session participants will be asked to report possible side effects occurring during tVNS and to rate their feeling on several visual analogue scales.
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tVNS — tVNS allows the non-invasive activation of the Vagus Nerve by delivering electrical pulses to the sensory afferent fibers of the auricular, thick-myelinated, branch of the vagus nerve in the outer ear. TVNS seems to engage the same neural pathways of invasive VNS methods and may provide a novel, bottom-up NIBS method to promote GABA release. tVNS will be performed by using a CE marked tVNS device. It consists in a programmable stimulation unit connected to two titan ear electrodes that are mounted on a gel frame, allowing to generate and transfer electric impulses from the stimulation unit to the surface of the skin, where the electrodes are applied.

SUMMARY:
The present study aims to assess the effects of non invasive electrical stimulation of the vagus nerve via transcutaneous vagus nerve stimulation (tVNS) on cognitive functions, inhibitory and tic control in patients with tic disorders. Taking into account the role that GABA plays in inhibitory control, the presence of alteration of GABA neurotransmission in Tic disorders and the possibility to increase GABA release with tVNS, the investigators hypothesized that tVNS might improve behavioral control in Tic disorders. Moreover, as suggested by previous studies investigating the effects of tVNS in other patient populations, the investigators expected that tVNS will be safe and well tolerated. Such results would encourage the use of tVNS in Tic disorders.

DETAILED DESCRIPTION:
The investigators planned a single centre, randomized, double-blind, sham- controlled, crossover (within subject) design.

Adults with Tic Disorders will be recruited and randomly assigned to two different groups: the active-tVNS group and the sham-tVNS group. Each group will undergo a two-sessions intervention during which active tVNS followed by sham tVNS or sham tVNS followed by active tVNS will be delivered in the active and sham tVNS group, respectively. The stimulation will be delivered during the execution of an inhibitory task and an attentional task. For the inhibitory task a Contextual Go No-Go paradigm will be used. During this task, participants will be presented with visual stimuli representing everyday actions embedded within congruent or incongruent context. For example, stimuli could consist in precision or grasping actions suggesting the intention to eat or to move the object in another place. For each stimulus, there will be a kinematic component consisting in the movement performed by the model and a contextual component, consisting in the embedding scenario of the action (a breakfast scenario, or a cleaning scenario). Participants will be instructed to press a button when a specific intention (go) will be suggested by the video and not to press a button for the opposite intention (no go), either according to the kinematics or to the context, depending on the experimental block. This way, it will be possible to assess inhibitory control at response level. Crucially, kinematics and context of the visual stimuli could point toward the same (congruent) or opposite (incongruent) intentions, thus allowing to assess inhibitory control at the stimulus level. For the attentional task, the attentional network test (ANT; Fan et al.,2002) will be used. The task is a modified version of a Flanker task and it allows measuring orienting, alerting and executive control components. To assess the clinical, neuropsychological and behavioural profiles, the Yale Global Tic Severity Rating Scale (YGTSS), the EuroQol quality of life questionnaire, the Raven Matrix, the Autism Quotient, the Barratt Impulsiveness scale and the Navon Task will be used. The effects of tVNS on patients' behavioural control (as assessed through the Contextual Go No-Go task and the ANT) will be related to clinical, neuropsychological and behavioural profile, for identifying best the features tVNS responder patients. Side effects will be tested after each session.

The protocol will allow testing the efficiency of tVNS in:

* enhancing inhibition at response level (response selection) in Tic disorders;
* enhancing inhibition at stimulus level (response inhibition) in Tic disorders;
* improving alerting, orienting or executive control in Tic disorders;
* improving patients' quality of life and Tic control;
* further investigating the safety and tolerability of tVNS.

ELIGIBILITY:
Inclusion Criteria:

* adults who aged 18-50 years;
* Diagnosis of Tic disorders

Exclusion Criteria:

* Presence of contraindication to tVNS (history of epilepsy in the last two years, severe brain trauma; presence of metal in the brain/skull or implanted neurostimulator, cardiac pacemaker; state of pregnancy);
* Recent changes in drugs therapy due to the intake of or the withdrawal from some drugs potentially changing the seizure threshold;
* Presence of comorbidity with an important medical condition;
* Severe sensorial, motor and/or behavioural problems that could interfere with the tasks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Contextual Go No-Go | Time 1- at the end the active session vs Time 0- at the end of the sham session
  Performance in the contextual go no go task, consisting in the accuracy in making the response in the presence of a go stimulus, and not responding in the presence of a no-go stimulus (Response selection) as a function of different level of congruency between the kinematics and the contextual cues (stimulus selection). Change in inhibition at response level (response selection) and at stimulus level (response inhibition) after active tVNS.
Attentional Network Test | Time 1- at the end the active session vs Time 0- at the end of the sham session
  Performance in the ANT tasks, with respect to the three components: alerting, orienting, executive control. For the alerting component, the mean RT of the correct trials in the double-cues conditions will be subtracted from the mean RT of the no-cue condition. For the Orienting component, the effect will be calculated by subtracting the mean RT of the spatial cue condition from the mean RT of the central cue condition. For the executive control component, the effect will be obtained by subtracting the mean RT of the incongruent flanking condition from the mean RT of the congruent flanking condition.Change in alerting, orienting, executive control after active tVNS.

SECONDARY OUTCOMES:
Tic control | Time 1- at the end the active tVNS session vs Time 0- at the end of the sham session
  Scores in the YBTCCS after each session will be compared.
tVNS feasibility | Time 1- at the end the active tVNS session vs Time 0- at the end of the sham session
  Evaluation of the number of dropouts: number of patients who renounce to complete the two sessions. Evaluation of the number of sessions completed per patient: total number of sessions performed in front of the total number proposed of two sessions
tVNS acceptability | Time 1- at the end the active tVNS session
  Ad-hoc questionnaire completed by participants to assess subjective evaluation of tVNS discomfort (10 cm Visual Analogue scales with higher values corresponding to greater discomfort).

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute, IRCCS E. Medea,, Pasian di Prato, Udine, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset will be availabe at https://osf.io/
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Before data analyses, for ten years.
Access Criteria: all
URL: https://osf.io/